CLINICAL TRIAL: NCT06898983
Title: Efficacy and Safety Study of Romiplostim N01 for Cancer Treatment-induced Thrombocytopenia (CTIT) in the Treatment of Leukemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Romiplostim N01-002
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Cancer Treatment-induced Thrombocytopenia (CTIT)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Romiplostim N01 (Experimental): Romiplostim N01 will be administered once weekly via subcutaneous injection upon the occurrence of Grade 3 thrombocytopenia (platelet count < 50×10⁹/L) following leukemia treatment. The recommended initial dose is 5 µg/kg, with a maximum single dose not exceeding 250 µg. A maximum of 8 doses may be administered during the treatment period.
  Interventions: Drug: Romiplostim N01

INTERVENTIONS:
Drug: Romiplostim N01 — Romiplostim N01 will be administered via subcutaneous injection once weekly when patients develop Grade 3 thrombocytopenia (platelet count < 50×10⁹/L) following leukemia treatment. The recommended initial dose is 5 µg/kg, with a maximum single dose not exceeding 250 µg. Treatment may continue for up to 8 doses.

SUMMARY:
Evaluation of the Efficacy and Safety of Romiplostim N01 for the Treatment of Cancer Treatment-Induced Thrombocytopenia (CTIT) in Patients with Leukemia

DETAILED DESCRIPTION:
Cancer treatment-induced thrombocytopenia (CTIT) refers to a decrease in platelet count caused by antitumor therapies during cancer treatment. It is a common adverse effect of anticancer treatment, with a particularly high incidence in patients with hematologic malignancies. CTIT increases the risk of bleeding, may limit treatment options, and can ultimately compromise the effectiveness of cancer therapy and reduce long-term survival. Currently, aside from platelet transfusion, thrombopoietic agents are commonly used to manage CTIT. Studies have shown that Romiplostim demonstrates a response rate of up to 71% in patients with chemotherapy-induced thrombocytopenia from solid tumors, with 89% of patients avoiding the need for platelet transfusion, thereby significantly reducing the risk of bleeding. However, there is limited evidence and a lack of prospective clinical trials investigating the use of Romiplostim in leukemia patients with CTIT. This study aims to evaluate the efficacy and safety of Romiplostim in adult leukemia patients with CTIT, in order to provide new therapeutic options and strategies, and ultimately improve the quality of life for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years, inclusive, regardless of sex;
* Histologically or pathologically confirmed diagnosis of leukemia;
* Patients with cancer treatment-induced thrombocytopenia (CTIT) in patients with leukemia due to antitumor therapy, with platelet count < 50×10⁹/L;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
* Subjects of childbearing potential agree to use reliable methods of contraception throughout the study period (including male or female condoms, contraceptive foam, gel, film, cream, suppository, abstinence, or intrauterine device);
* Patients considered by the investigator to potentially benefit from the study treatment;
* Voluntarily agrees to participate in the clinical trial, is fully informed of the study procedures, and has signed the written informed consent form.

Exclusion Criteria:

* Pregnant or breastfeeding women;
* Known hypersensitivity to Romiplostim N01;
* Presence of hematologic disorders other than cancer treatment-induced thrombocytopenia (CTIT) caused by leukemia treatment, including but not limited to primary immune thrombocytopenia, myeloproliferative disorders, multiple myeloma, or myelodysplastic syndromes;
* History of thrombocytopenia due to causes other than CTIT within 6 months prior to screening, including but not limited to chronic liver disease, hypersplenism, infections, or bleeding disorders;
* History of severe thrombotic events or known risk factors for thrombosis, or active thromboembolism requiring anticoagulation therapy;
* Severe bleeding within 2 weeks prior to screening (requiring more than 2 units of red blood cell transfusion or a sudden ≥10% drop in hematocrit);
* Use of thrombopoietin receptor agonists (e.g., eltrombopag), recombinant human thrombopoietin (rhTPO), or interleukin-11 (IL-11) within 1 month prior to screening;
* HIV infection;
* Chronic active hepatitis B or hepatitis C infection;
* Presence of severe infection or serious comorbidities involving the heart, liver, lungs, kidneys, nervous system, or metabolic diseases;
* Participation in any investigational drug or device clinical trial within 28 days prior to baseline visit;
* Subjects with cognitive impairment or uncontrolled psychiatric disorders;
* Refusal of the subject and/or legal representative to receive Romiplostim N01 treatment;
* Deemed unsuitable for enrollment by the investigator (e.g., comorbid conditions that may compromise subject safety or anticipated treatment non-adherence due to financial or other constraints).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Platelet response at Week 2 (PLT ≥ 50×10⁹/L) | 2 weeks
  Proportion of patients achieving a platelet count ≥ 50×10⁹/L at 2 weeks after initiation of treatment.

SECONDARY OUTCOMES:
Early Platelet Response Rate (within 7 days) | 7 days
  Proportion of patients achieving a response within 7 days of treatment initiation (Response defined as: no requirement for platelet transfusion and either a platelet count increase to ≥ 50×10⁹/L, at least a two-fold increase from baseline, or a platelet count ≥ 100×10⁹/L.)
Median time to platelet recovery without transfusion | 8 weeks
  Median time to achieve platelet counts of ≥ 50×10⁹/L and ≥ 100×10⁹/L without platelet transfusion.
Total platelet transfusion during treatment | 8 weeks
  Total platelet transfusion during treatment
Platelet nadir during treatment | 8 weeks
  Nadir platelet count during the treatment period (from initiation to end of treatment)

OTHER OUTCOMES:
Incidence of adverse events | Within 28 days after treatment discontinuation
  Incidence of adverse events
Incidence of bleeding events | Within 28 days after treatment discontinuation
  Incidence of bleeding events (based on World Health Organization bleeding assessment scale)
Survival outcomes | Within 28 days after treatment discontinuation
  Relapse-Free Survival (RFS), Overall Survival (OS), and Cumulative Incidence of Relapse (CIR)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Zhu, Ph.D, Principal Investigator — The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital)
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No